CLINICAL TRIAL: NCT00451529
Title: Predictive Value of Magnetic Resonance Imaging (MRI), 18-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET), and Microemboli Detection for Stroke
Brief Title: Predictive Value for Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dutch Heart Foundation (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Dr. M.E. Kooi, Dr. M.E. Kooi
Other Study IDs: 2006 B0
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with a moderate to severe carotid atherosclerotic plaque are at risk for stroke and this risk increases with increasing degree of stenosis. It has been shown that carotid endarterectomy in symptomatic patients with a carotid artery stenosis of 70-99% is highly beneficial. However, the beneficial effect of surgery in patients with symptomatic 30-69% stenosis is not clear yet.A clear beneficial effect of surgery in the 30-69% stenosis group might be found in a sub-group of patients whom are at greater risk for stroke. Definition of this sub-group might be achieved by plaque characterization, since rupture of a vulnerable plaque is the main cause of stroke due to carotid artery stenosis.This study will include patients with a 30-69% carotid artery stenosis, and assess plaque composition by MRI, the degree of plaque inflammation by FDG-PET, and the amount of microembolization by transcranial Doppler ultrasound. The main purpose of this study is to assess whether one or a combination of each of these imaging methods can predict the occurrence of a (recurrent) ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurological symptoms due to ischemia in the carotid artery territory and with a carotid stenosis between 30% and 69% as detected by ultrasound examination

Exclusion Criteria:

* Patients with a probable cardiac source of embolism (rhythm disorders, mitral valve stenosis, prolapse or calcification, mechanical cardiac valves, recent myocardial infarction, left ventricular thrombus, atrial myxoma, endocarditis, dilated cardiomyopathy, patent foramen ovale) or a clotting disorder.
* Patients with evident other cause of neurological symptoms than carotid stenosis due to atherosclerotic disease (like demyelinating diseases, epilepsy, congenital brain disorders, aneurysms, fibromuscular dysplasia, etc.).
* Patients already scheduled for carotid endarterectomy or stenting
* Severe co-morbidity, dementia, or pregnancy.
* Standard contra-indications for MRI (ferromagnetic implants like pacemakers or other electronic implants, metallic eye fragments, vascular clips, claustrophobia, documented allergy to contrast media, renal insufficiency, etc).
* Patients who were referred from another hospital to one of the three participating hospitals (to avoid referral bias).
* Patients who had a TIA or minor stroke more than 3 weeks before inclusion
* Patients who had a prior TIA or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of transient ischemic attack or minor stroke within three months of enrollment and an ipsilateral 30-69% carotid stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-08; Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne E Kooi, PhD, Principal Investigator — University Hospital Maastricht, Department of Radiology
Locations (1):
- University Hospital Maastricht, Department of Radiology, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Truijman MT, Kwee RM, van Hoof RH, Hermeling E, van Oostenbrugge RJ, Mess WH, Backes WH, Daemen MJ, Bucerius J, Wildberger JE, Kooi ME. Combined 18F-FDG PET-CT and DCE-MRI to assess inflammation and microvascularization in atherosclerotic plaques. Stroke. 2013 Dec;44(12):3568-70. doi: 10.1161/STROKEAHA.113.003140. Epub 2013 Oct 10. PMID 24114456